CLINICAL TRIAL: NCT00145886
Title: Effect of 12 Months Treatment With rhPTH on Calcium Balance, Bone Turnover, Bone Mineral Density, and Bone Micro-architecture in Patients With Fractures Associated With Low Bone Turnover and Sclerosing Bone Disorders
Brief Title: rhPTH Therapy for Low Turnover Bone Fragility
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12901A
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Osteopetrosis
Keywords: low bone turnover; sclerosing bone disorders,; osteopetrosis
MeSH Terms: conditions — Osteopetrosis | interventions — Parathyroid Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rhPTH (Experimental): Subjects will be treated rhPTH for 12 months
  Interventions: Drug: rhPTH

INTERVENTIONS:
Drug: rhPTH — Subjects will be treated with rhPTH for 12 months.
  Other Names: Recombinant Human Parathyroid Hormone

SUMMARY:
The purpose of this study is to determine how treatment with a new medication, recombinant human parathyroid hormone (rhPTH) affects calcium balance and bone strength.

DETAILED DESCRIPTION:
Subjects will have had a bone biopsy to definitively determine low bone turnover. Subjects and the treating doctor decide that treatment with rhPTH (recombinant human parathyroid hormone) is optimal before admission into the study. During the study, subjects will have several tests that will clarify how rhPTH is affecting calcium metabolism and bone properties. All of the studies will be performed in the University of Chicago General Clinical Research Center (GCRC).

To examine the effects of PTH (parathyroid hormone) on calcium metabolism, subjects will be admitted to the GCRC for 3 days in the beginning of the study. Subjects will have a plastic needle inserted into a vein to enable the nurses to draw your blood repeatedly without having to stick you every time. Subjects will have 120 mL (about 8 tablespoons) of blood drawn during the 3 day period. Subjects will be allowed to choose the food from the regular hospital menu but the amount of calcium from the diet will be the same during each day that you spend in the GCRC. The first day will be used to observe calcium balance without medication while the subsequent 2 days will be used to determine how calcium balance changes in response to the medication rhPTH. Subjects will take the medication in the morning, before breakfast - this will be considered time 0. During all 3 days, blood will be taken at 0, 2, 4, 6, 8, 12, 16, and 20 hours for examination of serum calcium and at 0, 4 and 12 hours for measurement of PTH (that is produced by your body).

On the first and 3rd day all the urine will be collected to measure how much calcium is lost in the urine.

After Subjects have received the medication for 3 months they will again be admitted to the GCRC, this time for 2 days during which they will continue to take the medication with the same measurements as on the last 2 days of the first admission. The same admission will be repeated after 12 months of treatment. During each of these admissions, you will have 80 mL (about 5 ½ tablespoons) of blood drawn.

In addition to these 3 inpatient stays in the CRC, subjects will also have several tests as an outpatient. The tests will be used to evaluate the effect of rhPTH on the bone. To this end, you will have 3 types of tests.

1. To evaluate the bone turnover (activity of bone cells) subjects will have blood and urine collected for measurement of biochemical markers of bone turnover (chemicals in the blood and urine that reflect the activity of bone cells) measured before and at 1, 2, 3, 6, 9, and 12 months. Subjects will have 10 mL (about 2 teaspoons) of blood drawn at each of these visits.
2. To evaluate changes in the bone density subjects will have bone density test of the lumbar spine, hip, heel and wrist measured every 3 months for 12 months.
3. To evaluate changes in the architecture or structure of the bone subjects will have 2 tests. First, the heel images that are obtained during the bone density test (under #2) will be subjected to radiographic texture analysis. This is a method of computerized analysis of the pattern of bone radiographic images which is supposed to differentiate between strong and weak bone based on the difference in the radiographic texture. The second test will be a bone biopsy. A bone biopsy involves inserting a needle through the skin and directly into the bone to obtain a piece of the bone of 1 cm (less than ½ inch) in length and 0.3 cm (1/10 inch) in diameter. Before this biopsy needle is inserted a numbing medication is injected to prevent pain during the procedure. You will also receive a medication through the vein so that you will be almost asleep during the procedure (intravenous sedation). Most people only experience minor pain for a few days after the biopsy. Subjects will have had the first bone biopsy before enrolling into this study. A second bone biopsy will be performed after 12 months of treatment with rhPTH.

ELIGIBILITY:
Inclusion Criteria:

* :patients with history of increased bone fragility by BMD criteria (T score > -1). In addition, the subjects will be enrolled only if they have clear evidence of low bone turnover as indicated by low normal levels of biochemical markers of bone turnover and finding of low bone turnover on bone biopsy. Each subject and his/her treating physician will have agreed that the rhPTH is the best treatment for the patient. Treatment with rhPTH will be considered only if the bone histomorphometry reveals a low turnover state and excludes other known forms of bone disease such as osteomalacia.

Exclusion Criteria:

* Subjects who are pregnant or younger than 20 will be excluded. Subjects cannot have osteoporosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2003-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To describe the acute effects of rhPTH administration on calcium balance. | The effects on calcium balance will be examined at the beginning, after 3 months, and after 12 months of treatment with rhPTH.
  The effects on calcium balance will be examined at the beginning, after 3 months, and after 12 months of treatment with rhPTH. The rational for examining calcium balance at these three time points is that (at least in patients wit osteoporosis treated with PTH) the initial response is primarily an increase in bone formation; at 3 months there is also a proportionate increase in bone resorption; and at 12 months there is an established general increase in bone turnover.

SECONDARY OUTCOMES:
To examine the effect of 12 months of therapy with rhPTH on bone density, bone turnover and bone micro-architecture. | Bone density will be measured at 0, 3, 6, and 12 months
  Bone density will be measured at 0, 3, 6, and 12 months in the lumbar spine, proximal femur, and distal radius using Lunar Prodigy, and in the calcaneus using Lunar PIXI (both from GE Medical Systems, Madison, Wisconsin).

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Vokes, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States